CLINICAL TRIAL: NCT03760393
Title: Using a Combined Health Action Process Approach and mHealth Intervention to Reduce Sedentary Behaviour in University Students - A Randomized Controlled Trial
Brief Title: A Combined HAPA and mHealth Intervention to Reduce Sedentary Behaviour in University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Dr. Harry Prapavessis, Professor, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HAPA Planning & SB in Students
Record Dates: First submitted 2018-11-24; First posted 2018-11-30 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Sedentary Lifestyle; Health Behaviour Change
Keywords: Sedentary Behaviour; Health Behaviour Change; Health Action Process Approach; mHealth; Intervention; Non-Sedentary Behaviours; Break Frequency; Break Duration; Action Planning; Coping Planning; Work Performance; Health Outcomes
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: This study will employ a prospective, 2-group, repeated measure (2x5), randomized controlled trial (RCT) design. All participants will be randomized into either a 6-week HAPA-treatment (SB-related planning + text messages intervention) or waitlisted control (no treatment) condition.
  All primary outcomes will be assessed at four time points (baseline, 2, 4, and 6 weeks), and again at a two-week follow-up (8 weeks). Action and coping planning and action control towards reducing occupational (student) sitting time will be assessed at the same time points. Secondary outcome assessments (i.e., work- and health-related outcomes) will occur pre-(baseline) and post-intervention (6 weeks).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HAPA-treatment (Experimental): (SB-related planning + daily text messages)
  Interventions: Behavioral: (SB-related planning + daily text messages)
- Control (No Intervention): (No Treatment) Participants randomly assigned to the control group will receive no information or intervention of any kind and will only be asked to complete the outcome questionnaires.

INTERVENTIONS:
Behavioral: (SB-related planning + daily text messages) — Participants will receive a one-on-one behavioral counseling session, and planning sheet as reference for developing strategies as part of their Action/Coping Plan. Participants will be asked to form 3-4 actions plans specifying when, where, how, and for how long they would reduce occupational (student) sitting time; and anticipate potential barriers and identify ways they could be overcome. Strategies will explicitly focus on the ultimate objective of increasing break frequency to every 30-45 minutes, achieving a break duration of 2-3 minutes, and increasing time spent standing and engaged in light-intensity PA, in the occupational domain (i.e. as a student; during school-related activities).
  Participants will also receive sedentary behaviour-related text messages twice daily, depending on their preferences and schedule, which will act as mini-booster interventions.
  Arms: HAPA-treatment

SUMMARY:
Societal changes have resulted in reduced demands to be active and increased daily time spent sitting. Sedentary behavior (SB) has been linked to many health problems such as type 2 diabetes and heart disease. University students are a high-risk population for excessive SB. Increasing the length and frequency of breaks from sitting and increasing the time spent standing and engaged in light physical activity are ways to decrease SB. The purpose of this study is to determine whether combining a Health Action Process Approach-based (theory-driven), specifically action and coping planning intervention, with a tailored text messaging intervention can reduce occupational (student) sitting time among university students. Participants in the intervention group will receive one behavioural counselling session, followed by daily, tailored text messages over a 6-week period, with a focus on encouraging them to reduce their sitting time as a student by increasing their frequency and duration of breaks from sitting, as well as time spent standing and engaged in light-intensity physical activity. It is expected that university students who receive the planning intervention and tailored text messages will report greater increases in non-sedentary behaviours (e.g., break frequency, break duration, standing, light physical activity) than those who do not receive the intervention.

DETAILED DESCRIPTION:
Using a randomized controlled trial design, the purpose of this study will be to examine whether combining a Health Action Process Approach (HAPA)-based intervention, specifically action and coping planning, with a tailored text message intervention can reduce occupational (student) sitting time by increasing frequency and length of breaks from sitting and non-exercise activity thermogenesis (NEAT) behaviours (i.e., standing, light-intensity physical activity) among university students. A secondary purpose will be to examine the effects of the intervention on participants' action planning, coping planning and action control regarding reducing their sitting time as a student, as well as self-rated work performance and health-related outcomes (i.e., role limitations due to physical health, role limitations due to personal or emotional problems, emotional well-being, and energy/fatigue). Another secondary objective will be to determine if action and coping planning and action control towards reducing occupational (student) sitting time are related to actual break behaviour, time spent standing, and time spent in light-intensity physical activity.

If successful, participants in the intervention group (sedentary intervention group) will report greater break frequency and break duration, time spent standing, and time spent in light-intensity physical activity, compared to participants in the control group (no treatment). In addition, it is hypothesized that participants in the intervention group will report greater action and coping planning and action control towards reducing sitting time as a student, as well as improved work- and health-related outcomes.

This study will employ a prospective, 2-group, repeated measure, randomized controlled trial (RCT) design. Participants will be full-time university and/or college students.

Potential participants (estimated enrolment: 112) will be recruited by Andrew Scott Rollo, Co-Investigator, for this study. Participants will be recruited from (1) undergraduate and graduate classes at the University of Western Ontario. Professors across faculties at UWO will be contacted via email and asked to (a) distribute the recruitment poster and study invitation to students in their course(s), and/or (b) allow study investigator(s) to provide a short presentation during their lecture time. The opportunity for students to participate will be posted on their UWO OWL site, as well as presented in their class. Participants will be instructed to contact the researcher via email and/or phone if they wish to participate or receive additional details prior to making a decision as to whether to participate. A second recruitment approach will involve recruiting full-time university and/or college students through recruitment posters distributed through social media (i.e., Facebook, LinkedIn). Recruitment posters and brief study details will be posted on social media. For social media outlets, permission from group administrators will be sought prior to posting social media recruitment materials, as applicable. As stated previous, university students interested in the study will be instructed to contact the researcher via email and/or phone to sign up for study participation.

At this point of contact, an email response will be sent to any interested individual. University students who choose to take part in this study will receive a link (with serial number authorization code) via email that directs them to the Letter of Information, electronic Informed Consent, and questionnaire for assessment of baseline measurements, which will be administered through a third party website called SoSci (online survey service). After viewing the Letter of Information and indicating that they consent to participate in the study (by clicking "I agree" on the survey), participants will be asked to complete a brief demographics questionnaire, followed by a questionnaire for baseline assessment of primary and secondary outcomes.

Upon completion of the Baseline assessment and prior to intervention delivery, all participants will be randomized, using computer-generated randomized stratification, into either a 6-week HAPA-treatment (SB-related planning + text messages intervention) or waitlisted control (no treatment) condition.

At this point, all participants will be sent a specific email (outlined below) depending on group assignment.

In the post-baseline questionnaire EMAIL response sent to intervention participants, participants (randomly assigned to the intervention group only) will be asked to provide a day and time (within 3 days of completing the baseline assessment) that they would be available to schedule the behavioural counselling session they will receive. As a follow-up to electronic consent, written consent will be obtained during administration of the behavioural counselling session.

In the post-baseline questionnaire EMAIL response sent to control participants, they will simply be reminded that they will receive a link to a questionnaire every two week for 8 weeks in their email and will be asked to complete these upon receiving them. Participants in the control group will also be asked to SIGN and RETURN the LOI/written informed consent via email at their earliest convenience.

For those in the treatment group, the study objective will be to reduce occupational (student) sitting time by increasing non- sedentary or NEAT behaviours (i.e., increasing break frequency to a break every 30-45 minutes, with each break having a duration of 2-4 minutes, and increasing their time spent standing and engaged in light- intensity PA. Participants randomly assigned to the control group will receive no information or intervention of any kind and will only be asked to complete the outcome questionnaires.

At the agreed upon and scheduled time, the researcher will deliver the intervention (i.e., implement the appropriate HAPA-based behavioural counselling session involving action and coping planning) either in person OR electronically via phone and an online presentation website (www.zoho.com) (only for those randomized into the intervention group). The method of delivery will entirely depend on the participant's availability, preference, and whether they live within driving distance of the investigator. To ensure equal numbers of local and remote participants, two computer-generated random number lists will be created by the lead investigator using an online research randomization program. Participants will be asked to complete a second informed consent (i.e., written informed consent) at this time.

The one-on-one counseling sessions will be delivered by the principal investigator to ensure standardization between participants. During the counseling session, the researcher will first ask if the participant has any strategies that he/she would like to try or think would be effective. As much as possible, strategies will be kept as original and specific to the participant's lifestyle as possible, while still fulfilling the study objectives. Upon creation of each strategy, the researcher will ask the participant if they think that the strategy they came up with is realistic. The number of strategies will also be personalized depending on how the participant's baseline measures compare to the objectives of their treatment group. This will be done in order to attenuate for any neglected/unused strategies by those with larger differences between baseline and objective values. Similarly, coping strategies will be created alongside each strategy in order to boost the adherence to the developed strategies. When an action plan strategy is developed, the researcher will ask the participant "what are some challenges you foresee with executing this strategy?", followed by "what do you think is something we can do in order to overcome this/these challenges?" This will be done in order to keep the coping strategies personalized to the participant's lifestyle. Overall, the behavioral counseling sessions will take approximately 20 minutes to complete. Participants will be given the form with their action plan and coping strategies and told to display it somewhere prominent so they will be reminded of the strategies. The principal investigator will conduct the planning interventions in a non-interfering manner by providing brief instructions and then remaining available to answer any questions.

All participants in the HAPA-treatment condition will then be entered into a contact list on the text-messaging website called "Oh Don't Forget." "Oh Don't Forget," is a Web-based application (http://ohdontforget.com) that works through "Recess Mobile" to send messages from a computer to mobile phone numbers that are programmed into the application. All participants will begin receiving tailored text messages the day after receiving their one-on-one counseling session. Every participant will receive the same daily texts as each other participant in their group, with times varying slightly depending on their schedule. As planning is an ongoing process, participants will be reminded (via text message) to formulate another set of action and coping plans at the beginning of weeks 3 and 5. Upon completion of the intervention period at 6 weeks, participants will be notified that they will no longer be receiving text messages and that the study is completed.

After the initial behavioural counseling session, ALL participants will be told they will receive a link to a questionnaire (assessment of primary and secondary outcomes) in their email every 2 weeks, for the next 6 weeks (i.e., weeks 2, 4, and 6), and to complete the questionnaire the day they receive it. Participants will also be told that 2 weeks following the end of the 6-week intervention, there will be a follow-up questionnaire (week 8), which they will receive and be asked to complete. Regardless of group assignment, all participants will complete the same outcome measures at Baseline, 2 weeks, 4 weeks, 6 weeks, and 2-week follow-up (8 weeks). All primary and secondary outcome questionnaires will be completed online and administered through a third party website called SoSci (online survey service). Participants in the HAPA-treatment condition will also be reminded via text to complete these.

The primary outcomes including frequency of breaks, length of breaks, and NEAT behaviours (i.e., standing, light- intensity PA) in the occupational domain of study (i.e., as a student) will be assessed using subjective, self-report approaches. Secondary analyses will be performed to examine effects of the intervention on theoretical determinants of behaviour change (i.e., action planning, coping planning, action control), as well as participants' perceived work-related outcomes (i.e., self-rated work performance) and health-related outcomes (i.e., role limitations due to physical health, role limitations due to personal or emotional problems, emotional well-being, and energy/fatigue). All primary outcomes will be assessed at four time points (baseline, 2, 4, and 6 weeks), and again at a two-week follow-up (8 weeks). Action and coping planning and action control towards reducing occupational (student) sitting time will be assessed at the same time points. Secondary outcome variables (i.e., perceived work- and health-related outcomes) will be assessed pre- (baseline) and post-intervention (6 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Must be 18+ years of age
* Must be a full-time university and/or college student
* Must be in self-reported good mental and physical health
* Must be able to read and write in English
* Must have access to a computer with Internet
* Must own a mobile phone with free unlimited incoming text messages.

Exclusion Criteria:

* Under 18 years of age
* Do not read or write in English
* Not a full-time university and/or college student
* Do not have access to a computer with Internet
* Do not own a mobile phone with free unlimited incoming text messages and/or emails
* Pregnant
* Medical condition that prohibits individual from being physically active.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Changes in Frequency of Breaks from Sitting as a Student | Baseline, Weeks 2, 4, 6, and at the 2-week follow-up (Week 8)
  Modified version of the SIT-Q 7d (Wijndaele et al., 2014; Sui & Prapavessis, 2016); 1-item; 12-point scale (Less than every 30 min, Every 30-45 min, Every 45 min-1 hour, Every 1-1.5 hours, Every 1.5-2 hours, Every 2-3 hours, Every 3-4 hours, Every 4-5 hours, Over every 5 hours, No interruption). Lower values represent a better outcome.
Changes in Duration of Breaks from Sitting as a Student | Baseline, Weeks 2, 4, 6, and at the 2-week follow-up (Week 8)
  Modified version of the SIT-Q 7d (Wijndaele et al., 2014; Sui & Prapavessis, 2016); 1-item; 10-point scale (Less than 30 sec, 30 sec-1 min, 1-2 min, 2-3 min, 3-4 min, 4-5 min, 5-10 min, 10-15 min, 15-30 min, Over 30 min). Higher values represent a better outcome.
Changes in Time Spent Standing as a Student | Baseline, Weeks 2, 4, 6, and at the 2-week follow-up (Week 8)
  Five-item modified Occupational Sitting and Physical Activity Questionnaire (OSPAQ; Chau, Van Der Ploeg, Dunn, Kurko, & Bauman, 2012)
Changes in Time Spent Engaged in Light-Intensity Physical Activity (i.e., walking) as a Student | Baseline, Weeks 2, 4, 6, and at the 2-week follow-up (Week 8)
  Five-item modified Occupational Sitting and Physical Activity Questionnaire (OSPAQ; Chau, Van Der Ploeg, Dunn, Kurko, & Bauman, 2012)

SECONDARY OUTCOMES:
Action Planning towards reducing occupational (student) sitting time | Baseline, Weeks 2, 4, 6, and at the 2-week follow-up (Week 8)
  Four-items; five-point Likert scale (1 = "completely disagree" to 5 = "totally agree")
Coping Planning towards reducing occupational (student) sitting time | Baseline, Weeks 2, 4, 6, and at the 2-week follow-up (Week 8)
  Five-items; five-point Likert scale (1 = "completely disagree" to 5 = "totally agree")
Action Control towards reducing occupational (student) sitting time | Baseline, Weeks 2, 4, 6, and at the 2-week follow-up (Week 8)
  Six-items; five-point Likert scale (1 = "completely disagree" to 5 = "totally agree")
Self-rated Work Performance | Baseline, Week 6
  One-item, 11-point Likert scale (0-10; 0 = Absolutely unacceptable, 10 = Absolutely Ideal). Higher values represent a better outcome.
Role limitations due to physical health | Baseline, Week 6
  RAND 36-item Short Form Survey (SF-36; Ware and Sherbourne, 1992) modified version (16-item). Four-items will assess participant's perceived role limitations due to physical health problems; 2-point scale (yes, no)
Role limitations due to emotional health | Baseline, Week 6
  RAND 36-item Short Form Survey (SF-36; Ware and Sherbourne, 1992) modified version (16-item). Three-items will assess role limitations due to personal or emotional problems; 2-point scale (yes, no)
Emotional well-being | Baseline, Week 6
  RAND 36-item Short Form Survey (SF-36; Ware and Sherbourne, 1992) modified version (16-item). Five-items will assess perceived emotional well-being; 5-point Likert scale (All of the time =1, Most of the time = 2, Some of the time = 3, A little of the time = 4, None of the time = 5)
Energy/Fatigue | Baseline, Week 6
  RAND 36-item Short Form Survey (SF-36; Ware and Sherbourne, 1992) modified version (16-item). Four-items will assess perceived energy/fatigue; 5-point Likert scale (All of the time =1, Most of the time = 2, Some of the time = 3, A little of the time = 4, None of the time = 5)

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Western Ontario, London, Ontario, Canada